CLINICAL TRIAL: NCT02178566
Title: Pulmonary Rehabilitation in COPD: Response to Inhaled Treprostinil (Tyvaso)
Brief Title: Pulmonary Rehab in Chronic Obstructive Pulmonary Disease (COPD): Response to Tyvaso
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to enroll
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Inova-TY-PR-001
Record Dates: First submitted 2014-06-22; First posted 2014-07-01 (Estimated); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Trepostinil; Pulmonary Rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — treprostinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled Treprostinil Placebo (Placebo Comparator): A dose of placebo resembling inhaled treprostinil will be administered to all study participants in the placebo comparator arm prior to each of their Pulmonary Rehab sessions. A dose of inhaled albuterol will be administered prior to each inhaled agent. Vitals signs will be taken prior to administering the dose and no medication will be given if the systolic blood pressure in < 85 mm Hg. Three puffs of inhaled trepostinil dose will be administered each time to all patients .
  Interventions: Drug: Inhaled Treprostinil
- Inhaled Treprostinil (Active Comparator): A dose of inhaled treprostinil will be administered to all study participants prior to each of their Pulmonary Rehab sessions. A dose of inhaled albuterol will be administered prior to each inhaled agent. Vitals signs will be taken prior to administering the dose and no medication will be given if the systolic blood pressure in < 85 mm Hg. Three puffs of inhaled treprostinil dose will be administered each time to all patients .
  Interventions: Drug: Inhaled Treprostinil

INTERVENTIONS:
Drug: Inhaled Treprostinil — A dose of inhaled treprostinil or placebo will be administered to all study participants prior to each of their Pulmonary Rehab sessions. Three puffs of inhaled treprostinil dose will be administered each time to all patients .
  Other Names: Tyvaso

SUMMARY:
The investigators' hypothesis is that pretreating patients with COPD with inhaled treprostinil prior to pulmonary rehabilitation sessions will result in improved exercise tolerance during sessions. This in turn will lead to an increased response to pulmonary rehabilitation, resulting in improved exercise tolerance and quality of life.

DETAILED DESCRIPTION:
Study Hypothesis:

Our hypothesis is that pre-treating patients with COPD with inhaled treprostinil prior to pulmonary rehabilitation sessions will result in improved exercise tolerance during sessions. This in turn will lead to an increased response to pulmonary rehabilitation, resulting in improved exercise tolerance and quality of life.

Study Background:

Pulmonary rehabilitation (PR) is a widely accepted intervention in patients with advanced COPD. This has consistently been shown to improve patients' quality of life and functional ability. Indeed, enrollment and completion of a course of PR is a prerequisite prior to major interventions such as lung volume reduction surgery or transplantation. A typical course of PR includes 20 sessions of supervised exercise and educational activity over an 8 week period. Sessions are usually held three times per week and last between 2-3 hours each. Most patients with COPD will have a ventilatory limitation to exercise and while many are oxygen dependent, a minority of patients will have a true hypoxic limitation to exercise. Nonetheless, when patients with COPD are ambulated on oxygen they feel better and walk further. Indeed, supplemental oxygen remains one of the few interventions that have been demonstrated to be associated with improved survival in patients with COPD.

There have been a few studies and case reports utilizing inhaled pulmonary vasodilators in patients with COPD, although none to date have used treprostinil. One study of 10 patients with COPD and pulmonary hypertension found improved gas exchange and exercise tolerance following using of inhaled iloprost an alternative inhaled pulmonary vasodilator. No adverse effects were observed. [Dernaika TA, Beavin M, Kinasewitz GT. Iloprost improves gas exchange and exercise tolerance in patients with pulmonary hypertension and chronic obstructive pulmonary disease. Respiration; 2010: 79(5): 377-382.)] A case report of a patient with pulmonary hypertension and COPD found sustained improvements in exercise tolerance with regular use of inhaled iloprost. [Hegewald MJ, Elliott CG. Sustained improvement with iloprost in a COPD patient with severe pulmonary hypertension. Chest 2009; 135(2): 536-537.] While these limited trials support the concept of physiologic improvement with use of inhaled pulmonary vasodilators in COPD, our study differs from these in several important ways. This study is unique in that there has never been a prior similar study of medication pretreatment prior to PR to enhance exercise performance in any patient subgroup. Furthermore, treprostinil has not yet been evaluated for use on an as needed basis.

Indication Studied:

COPD/Pulmonary rehabilitation

Study Objectives:

* Primary Objective: To determine the effect of inhaled treprostinil, administered prior to pulmonary rehabilitation sessions, on the six minute walk test distance (6MWT) in COPD patients after completing an 8 week course of pulmonary rehabilitation
* Secondary Objectives: To assess the effect inhaled treprostinil, administered prior to pulmonary rehabilitation in COPD patients, on secondary outcomes including quality of life (as measured by the St. George's respiratory questionnaire, Clinical COPD Questionaire), BODE index, lowest nadir of oxygen saturation on 6 minute walk test, number of exacerbations, ER visits, hospitalizations, and change in measures of strength training.

Trial Design:

An adaptive, prospective, randomized, double-blind, placebo-controlled study of 34 patients with advanced COPD who have been referred for pulmonary rehabilitation. All patients will be screened at baseline with an arterial blood gas. A test dose of inhaled nitric oxide (NO) will be administered to all subjects for 2-5 minutes. An ABG will then be repeated. Patients who have a worsened A-a gradient will be screened out. Patients will be randomized to receive one dose of inhaled treprostinil or placebo prior to each of their exercise sessions. All patients will be pretreated with albuterol prior to the dose of inhaled treprostinil (or placebo).

Patient Population:

We plan to screen 50 patients with a goal of enrolling 34 patients. Patients referred for pulmonary rehabilitation at Inova Fairfax Hospital with moderate to severe COPD as a primary diagnosis will be screened for inclusion in the trial. Inclusion and exclusion criteria are listed below.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign informed consent prior to initiation of any study mandated procedure
2. Male or female ≥ 40 years of age
3. Women of childbearing potential must use a reliable method of contraception from screening until 1 month after end of study medication
4. Clinical diagnosis of moderate to severe COPD, with an obstructive pattern on pulmonary function tests showing both:

   * FEV1/FVC < 0.7 and
   * FEV1 ≤ 60% of predicted value, on standard COPD therapy
5. Current or past smokers of ≥ 10 pack years
6. If taking oral (< 20 mg/day of prednisone equivalent) or inhaled corticosteroids, inhaled beta-agonists (short and long acting), or inhaled muscarinic antagonists (short and long acting), or statins the dose must be stable for at least 30 days prior to initial PR visit.
7. Ability to adequately participate in exercise testing/pulmonary rehabilitation program with supplemental oxygen use over the period of the study (in the best opinion of the investigator)

Exclusion Criteria:

1. Patients fulfilling one or more of the following criteria of documented COPD exacerbation within 1 months prior to screening:

   * Use of antibiotics for COPD exacerbation
   * Initiation or dose increase of steroids (inhaled, oral or intravenous) for COPD exacerbation
   * Hospitalization for COPD exacerbation
2. BMI > 40 kg/m2
3. Unstable coronary artery disease, unstable angina, or myocardial infarction within 3 months prior to screening
4. History of pulmonary edema, or uncontrolled heart failure
5. Uncontrolled systemic hypertension with a blood pressure >180/105 mmHg at rest
6. Systemic hypotension with systolic blood pressure < 85 mmHg
7. Uncontrolled arrhythmias
8. History of syncope
9. Planned surgical intervention during the study period
10. Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results including musculo-skeletal limitations, peripheral arterial disease, drug or alcohol dependence or psychiatric disease
11. Severe hepatic impairment (Child-Pugh Class C)
12. Chronic renal insufficiency, as defined by serum creatinine of > 2.5 mg/dL or estimated creatinine clearance < 30 mL/min or the requirement for dialysis
13. Pregnant or nursing
14. Currently (within 30 days prior to enrollment) taking specific pulmonary arterial hypertension therapy (e.g., bosentan, ambrisentan, tadalafil, sildenafil, epoprostenol, treprostinil, iloprost, beraprost), sildenafil and tadalafil for erectile dysfunction is permitted
15. Initiation of a pulmonary rehabilitation program within 3 months prior to screening or initiation or changes during the study
16. Participation in any other clinical trial, except observational, or receipt of an investigational medicinal product within 30 days prior to RHC visit
17. Known concomitant life-threatening disease with a life expectancy < 6 months
18. Known hypersensitivity to treprostinil or any of the excipients of the drug formulations.
19. Known hypersensitivity to inhaled nitric oxide

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Nathan, MD, Principal Investigator — Inova Fairfax Medical Campus; Christopher King, MD, Principal Investigator — Inova Fairfax Medical Campus
Locations (1):
- Inova Fairfax Medical Campus, Falls Church, Virginia, United States

REFERENCES:
- [Background] Dernaika TA, Beavin M, Kinasewitz GT. Iloprost improves gas exchange and exercise tolerance in patients with pulmonary hypertension and chronic obstructive pulmonary disease. Respiration. 2010;79(5):377-82. doi: 10.1159/000242498. Epub 2009 Sep 25. PMID 19786728
- [Background] Hegewald MJ, Elliott CG. Sustained improvement with iloprost in a COPD patient with severe pulmonary hypertension. Chest. 2009 Feb;135(2):536-537. doi: 10.1378/chest.08-1515. PMID 19201716

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Inhaled Treprostinil Placebo | Inhaled Treprostinil
Started (no data available) | 0 | 1 (no data available)
Completed (no data available) | 0 | 0 (no data available)
Not Completed | 0 | 1
Not completed — patient did not complete due to noncompliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 patient enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Treprostinil Placebo | Inhaled Treprostinil | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 61 | 61 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 1 | 1
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Distance Walked on 6MWT
Description: To determine the effect of inhaled treprostinil, administered prior to pulmonary rehabilitation sessions, on the six minute walk test distance (6MWT) in COPD patients after completing an 8 week course of pulmonary rehabilitation
Time Frame: 9 weeks
Population: no patient completed. one patient consented but did not complete the study
Groups:
- Inhaled Treprostinil Placebo: A dose of placebo resembling inhaled treprostinil will be administered to all study participants in the placebo comparator arm prior to each of their Pulmonary Rehab sessions. A dose of inhaled albuterol will be administered prior to each inhaled agent. Vitals signs will be taken prior to administering the dose and no medication will be given if the systolic blood pressure in < 85 mm Hg. Three puffs of inhaled trepostinil dose will be administered each time to all patients .
  No patient completed
- Inhaled Treprostinil: A dose of inhaled treprostinil will be administered to all study participants prior to each of their Pulmonary Rehab sessions. A dose of inhaled albuterol will be administered prior to each inhaled agent. Vitals signs will be taken prior to administering the dose and no medication will be given if the systolic blood pressure in < 85 mm Hg. Three puffs of inhaled treprostinil dose will be administered each time to all patients .
  no patient completed
Arm/Group | Inhaled Treprostinil Placebo | Inhaled Treprostinil
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Patients monitored from dosing to end of study treatment period.
Arm/Group | Inhaled Treprostinil Placebo | Inhaled Treprostinil
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Treprostinil Placebo (N=0) | Inhaled Treprostinil (N=1)
Lightheadedness (General disorders) | 0 (0) | 1 (2) — Patient reported jittery feeling and lightheadedness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT02178566/Prot_SAP_000.pdf